CLINICAL TRIAL: NCT00114322
Title: Comparing Wavelengths Using LED Light for SAD Treatment
Brief Title: Light-Emitting Diode (LED) Light for Seasonal Affective Disorder (SAD) Treatment
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Brigham and Women's Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2005-P-000160
Record Dates: First submitted 2005-06-14; First posted 2005-06-15 (Estimated); Last update posted 2007-01-15 (Estimated); Status verified 2005-06

CONDITIONS: Seasonal Affective Disorder
MeSH Terms: conditions — Seasonal Affective Disorder

INTERVENTIONS:
Device: light exposure from LED source at narrow 468 nm or broader 400-700 nm wavelength

SUMMARY:
Recurrent fall/winter major depression (known as Seasonal Affective Disorder (SAD)) is a prevalent and disruptive disorder whose pathophysiological basis is unknown, but several hypotheses attribute a causal role to the circadian timing system. Bright white light exposure via the retina has been shown to reverse the symptoms of SAD. Recent physiological studies demonstrated the existence of retinal ganglion cells capable of transducing light input to the retinohypothalamic tract, the primary circadian afferent in humans. This retinohypothalamic system appears to be maximally sensitive to light in the 446-477nm (violet/blue) range.

Using light-emitting diode (LED) technology, light of narrow bandwidths now can be delivered from a safe, relatively inexpensive device. We propose to contrast in SAD patients the efficacy and tolerability of 468 nm LED light from a portable 11cm x 6cm commercially-available device (GoLITEÔ) to a broader 400-700 nm wavelength LED-generated light housed in an identical device. The broad wavelength (white) light from our LED device is similar to that from cool-white fluorescent 10,000 lux devices currently the standard for treatment of SAD (see e.g., Lam & Levitt, 1999).

Twenty-four depressed SAD outpatients will be randomized to a 3-week trial of light therapy using either the narrow 468 nm LED source or the broader 400-700 nm LED source, each housed in a GoLITEÔ device. Subjects will be given devices and written instruction for administering daily treatments at home, 45min every (q) a.m. The devices will be described to subjects in terms of wavelength but not specifically described as "blue" or "white." Weekly depression ratings and assessments of adverse effects will be obtained by a trained rater blind to the treatment condition. Depressive symptoms will be rated weekly by the same trained clinician.

The following hypotheses will be evaluated:

* H1-- Depressed SAD patients will demonstrate greater antidepressant therapeutic benefit from the narrow-wavelength (blue) source than from the broad-wavelength (white) source.
* H2-- Depressed SAD patients will manifest fewer adverse effects during treatment with the narrow-wavelength (blue) source than with the broad-wavelength (white) source.

DETAILED DESCRIPTION:
BACKGROUND AND SIGNIFICANCE

Discovery in the late 1970s that bright light affects neuroendocrine rhythms such as melatonin secretion, and can reset the circadian pacemaker in humans, paved the way for the discovery that seasonally recurrent fall/winter depressions--christened Seasonal Affective Disorder (SAD)--can be treated with bright light exposure (Lewy et al., 1980; Rosenthal et al., 1985). It was reasoned that seasonal rhythms of mood in humans, like other seasonal physiological cycles in mammals, could be regulated by the biological "clock." A series of studies has demonstrated that bright light exposure does produce therapeutic effects in SAD patients beyond the level achieved by placebos (Eastman et al., 1998; Lewy et al., 1998; Terman et al., 1998) and that retinal exposure is required for efficacious treatment (Wehr et al., 1987; Koorengevel, 2001).

Attempts to construct an action spectrum for suppression of melatonin secretion and for resetting the circadian pacemaker suggest that 446-477 nm wavelengths are most potent (Brainard et al., 2001; Lockley et al., 2003), which is inconsistent with rod or cone mediation of the responses (Brainard, 2004). Discovery that a melanopsin-containing system of retinal ganglion cells serves as a primary afferent to the hypothalamic circadian pacemaker (Provencio et al., 2000; Gooley et al, 2001; Hattar et al, 2002) suggests a possible basis for the potency of violet/blue light on these neuroendocrine circadian endpoints and raises the possibility that light of this wavelength also might be uniquely potent for treatment of SAD (Brainard, 2004).

Estimates of SAD prevalence range from 0.4 - 9.7% of the general population in the United States, depending on the survey methods and precise criteria used (Rosen et al., 1990; Blazer et al., 1998). In addition to those with recurrent episodes of frank Major Depression, patients with less severe "sub-syndromal" winter depression and those with annual exacerbation of a year-round mood disorder also have been shown to benefit from light treatment in fall/winter months (Kasper et al., 1989). Since the 1990s, cool-white fluorescent sources capable of yielding 10,000 lux polychromatic white light have been the treatment standard (Lewy et al., 1998; Terman et al., 1998; Desan et al., 2001; also see e.g., Lam & Levitt, 1999). Although well-tolerated, some transient adverse effects of the 10,000 lux white light have been reported, such as agitation or feeling "wired," insomnia, headache, eye or vision problems, nausea, sedation, and chest tightness (Labbate et al., 1994; Kogan et al., 1998; Terman & Terman, 1999). The more common of these complaints--headache, eye or vision problems, and insomnia--remit rapidly after discontinuation of light exposure (Oren et al., 1991), however, narrower bandwidth light if more potent in antidepressant effectiveness might be administered at lower intensities and thereby further reduce adverse effects and increase tolerability of the treatment (Brainard, 2004).

A between-subjects double-blind comparison of 3-weeks treatment using narrow-band LED panels at blue (468 nm at 500 mW/cm2) vs red (700 nm at 15 mW/cm2) wavelengths in 24 SAD patients demonstrated both greater reductions in depressive symptoms and also remission rates (54.5% vs 30.8%) in favor of the blue light source (Byrne et al., 2004). Comparisons of this narrow bandwidth blue LED light with white light would be of even greater clinical interest since white fluorescent sources currently are the industry standard.

Safety

At the irradiance levels emitted by commonly utilized light therapy devices, dermatologic safety concerns are minimal. Similarly, thermal damage to cornea, lens or retina requires milliwatt-to-watt exposure, far in excess of that emitted from the therapeutic devices. Ocular safety for 10,000 lux white fluorescent sources has been assessed and comprehensive ophthalmologic examinations of individuals with healthy eyes who used white-light therapy daily during fall/winter months for up to 5 years did not reveal adverse effects (Gallin et al., 1995; Gorman et al., 1993). Shorter wavelengths of light are of greater concern due to photo-keratitis of the cornea and cataract of the lens from 180-400nm ultraviolet light, and photochemical injury to the retina at 310-550 nm with a peak near 440 nm (Sliney, 2004). The blue-light LED source to be utilized in the present research (Go-LITE™) was determined to have an averaged radiance well below the 10-mW/cm2*sr safety limit for continuous viewing.

RECRUITMENT PROCEDURES

We will recruit adults, age 18-64 years, who meet diagnostic criteria for seasonal affective disorder by means of public service announcements in the community. The approved announcement will be released via the Partners weekly research announcement system, may be disseminated to press outlets, and will be used on the voice mail menu of Dr. Anderson's SAD clinical services at BWH. An informational webpage linked to the BWH website (http://www.brighamandwomens.org/psychiatry/Research/sadresearch.asp) will provide more detailed information and a mechanism for prospective subjects to request further information. Interested individuals will be directed to a research assistant at the BWH Clinical Trials Center who will answer questions regarding the study and will conduct a telephone screening to assess eligibility. Those subjects found eligible and interested will be referred by the research assistant for a psychological screening interview.

CONSENT PROCEDURES

Each subject will be enrolled by his or her written informed consent obtained by members of the study staff. Following an initial telephone screening, each prospective subject will undergo an in-depth psychological evaluation at BWH by the principal investigator, Janis L. Anderson, PhD., or at McLean Hospital by Carol Glod, RN, Ph.D. Prior to the psychological screening, Dr. Anderson or Dr. Glod will review the Screening Consent Form with the subject. Dr. Anderson is an experienced clinical psychologist and Dr. Glod is an experienced doctor of nursing; each is trained to consider both cognitive and emotional factors that affect the ability to consent. If written informed consent is obtained on the Screening Consent Form then the psychological evaluation will take place. In that evaluation meeting, Dr. Anderson or Dr. Glod also will present the subject with a copy of the Study Consent Form to review and take home. Subjects will be encouraged to inform their medical providers and therapists about their interest in participating in the study. The meetings with Dr. Anderson or Dr. Glod will be scheduled in advance; nothing in the circumstances of this protocol would require a hasty decision on the part of the potential subject. Subsequent to the psychological screening for prospective subjects who meet diagnostic criteria, a medical examination will be performed by a doctor of Ophthalmology. If the subject is found to meet all inclusion criteria for the study, doctor of Ophthalmology, a licensed physician, will review the Study Consent Form and obtain written informed consent for the study procedures themselves. Upon each outpatient visit for the study procedures, the subject's mental status will be reassessed. However, due to the nature of SAD symptoms and the inclusion/exclusion criteria for the present study, we do not anticipate enrolling subjects whose ability to consent would be transitory.

RESEARCH DESIGN AND METHODS

A between-subjects double-blind trial will compare daily outpatient treatment using a narrow (468 nm, 27 nm half-peak bandwidth) LED light source (GoLITE™) to a broad 400-700 nm wavelength LED-generated light housed in an identical device in 24 seasonally-depressed adults. Dependent variables will be severity of depression and extent of adverse effects.

Research procedures will not begin in the Autumn/Winter until the subject has a depression rating of at least 20 on the SIGH-SAD (Structured Interview Guide for the Hamilton Depression Rating Scale-Seasonal Affective Disorders Version; Williams et al., 1988). The SIGH-SAD is a structured clinical interview for rating not only the traditional Hamilton Depression Rating Scale items but also the "atypical" vegetative symptoms characteristic of SAD. The validity of and reliability of the SIGH-SAD is well-established, and it is the preferred instrument for assessing symptom severity in SAD studies (e.g., see Lam & Levitt, 1999). A companion instrument, the Hypomania Interview Guide for Seasonal Affective Disorder (HIGH-SAD) also will be administered. A rater, who will be blind to the treatment condition of the subjects, will administer the SIGH-SAD and HIGH-SAD prior to and for each week during the 3-wk trial.

Subjects will begin treatment when post-treatment SIGH-SAD depression score ≥ 20. Dr. Anderson or Dr. Glod will meet with each subject to provide the light device and instruction for its outpatient use as detailed below. The subject will be asked to sign a written agreement for return of the light device. Subjects will use the light device and return weekly for symptom ratings; each will be seen by Dr. Anderson or Dr. Glod as well. At the conclusion of the 3-wk trial, Dr. Anderson or Dr. Glod will meet with the subject to discuss their response to light treatment and the indications for continuing light treatment through the end of that winter. Subjects will be offered the opportunity to keep the same device or try the other device until the end of the fall/winter season and will be followed monthly if they choose to do so. Alternative treatment modalities also will be discussed and referrals for follow-up care provided as indicated. All forms of SAD treatment will cease by June 1.

EQUITABLE SELECTION OF SUBJECTS

SAD is diagnosed on the basis of history and a definitive diagnosis is difficult to make in adolescents. In addition, their symptom profile differs from that seen in adults which would make assessment using any single measure difficult and would require a substantially larger sample size. Therefore in this preliminary investigation we propose to recruit individuals between the ages of 18-64. Because the safety of light treatment in pregnancy has not been established, and because mood effects of pregnancy and recent delivery would complicate assessment of treatment response in this 3-wk trial, only nonpregnant, non-lactating women will be included.

Recruitment will be by public means and no one will be excluded on the basis of race, gender, ethnic background, or other demographic factors. Dr. Anderson is responsible for outpatient monitoring of light treatment and is only fluent in English. Therefore, if potential subjects do not understand English it will be necessary to have available a bilingual physician in the community who would be able to work with Dr. Anderson in providing outpatient care.

PRIVACY AND CONFIDENTIALITY

Disclosure of Information Outside Partners:

Identifying information will be recorded only on screening contact sheets (which will be maintained under secure conditions in the Clinical Trials Center and later stored in locking file cabinets in a locked research room at 221 Longwood Ave. under the control of Dr. Anderson), on the signed consent forms (stored in locking file cabinets in a locked research room at 221 Longwood Ave. under the control of Dr. Anderson or at McLean Hospital under the control of Dr. Glod), and in emails sent within the Partners system to staff members who schedule the appointments, obtain laboratory specimen; or conduct symptom ratings.

All data will be stored in computer files with code number for the subjects; no identifiers other than the code number will be kept in the data files nor will they be used in any reports or publications concerning this research. The key for the code will be kept in locking file cabinets in a locked research room at 221 Longwood Ave. under the control of Dr. Anderson or at McLean Hospital under the control of Dr. Glod.

Any records that may be of use to other treatment providers for purposes of continuity of care, whether at Partners institutions or elsewhere, will be released upon written authorization of the subject or their legal representative in accordance with current applicable laws and regulations.

EXPECTED BENEFITS

Patients with seasonal affective disorder may experience relief from symptoms with light therapy during this study. If the treatment is effective, they may continue it with equipment from and supervision by Dr. Anderson or Dr. Glod through the end of the winter season. If the treatment is not effective, referrals for additional treatment will be made. However, relief from depression is in no way guaranteed.

FORESEEABLE RISKS AND DISCOMFORTS

1. Blood drawing. There may be some discomfort or bruising on initial insertion into a vein. There is a rare possibility of developing a small blood clot, inflammation, or local infection. Fainting may rarely occur in individuals very uncomfortable with blood drawing procedures.
2. Light treatment. Safety of equipment. Light therapy with bright fluorescent light has been tested in many individuals and serious irreversible adverse effects have not been reported. The most common side effect of light therapy is irritability or agitation that remits after termination of the light or decrease of the daily duration of exposure. Participants will be carefully monitored for such side effects and light therapy exposure will be decreased or eliminated if these adverse effects occur. Although light treatment has been tested in pregnant women in a small number of studies, the safety of light treatment in pregnant women has not been conclusively established. Female subjects will be told that participation in this study may be hazardous to an embryo or fetus and therefore that it is essential that adequate birth control be used while participating. If they should become pregnant while in the study, they should notify the investigators immediately.

MINIMIZATION OF RISKS AND SAFETY MONITORING

Subjects will be instructed to begin daily 45-min sessions of exposure to the light each morning shortly after they awaken (provided it is after 6 a.m.). Written instructions will be given, potential adverse effects will be discussed, and subjects will be instructed to telephone the supervising clinician (either Dr. Anderson or Dr. Glod) with any questions or should any adverse effects occur. A telephone appointment will be scheduled for 2-3 days after the first use of the light device. Patients who complain of feelings of jitteriness after using the light device will be advised to reduce their duration of daily exposure to 30 min per day. Patients who complain of headache after using the light device each day for 2-3 days will be advised to return for a visit to review the procedures they are using. An appointment will be scheduled for 7 days after the first use of the light device. Any patient who continues to complain of headache after the first week of light exposure will be withdrawn from the study. Patients who complain of feelings of jitteriness after using the light device 20 min per day will be withdrawn from the study.

An appointment will be scheduled for 14 days and 21 days after the first use of the light device. In general, the criteria for withdrawing patients from the study are based on Axis V of the DSM-IV, Global Assessment of Functioning (GAF). No patient with a GAF less than 50 will be enrolled in this study, and any patient whose GAF decreases to less than 50 during the course of the study will be withdrawn. This specifically includes, but is not limited to, any patient reporting suicidal ideation, symptoms of psychosis, or symptoms of mania at any point during the study will be withdrawn from the study and evaluated immediately by Dr. Anderson or Dr. Glod for treatment.

Any adverse events will be reported promptly to the Human Research Committee.

ELIGIBILITY:
Inclusion Criteria:

* History of recurrent major depressive episodes with winter-type seasonal pattern by Diagnostic and Statistical Manual of the American Psychiatric Association, 4th Ed. (DSM-IV) criteria (American Psychiatric Association, 1990), based on diagnostic interview utilizing the Structured Clinical Interview for DSM-IV Axis I Disorders (SCID) and graphic diagnostic tool
* Free of medical illness, not pregnant, as determined by detailed history and physical examination including blood and urine chemistries and thyroid function tests

Exclusion Criteria:

* History of concurrent psychiatric illness that would preclude compliance with the protocol and ability to complete the study safely
* Active suicidal or homicidal ideation or plan
* Variable psychiatric symptoms such as rapid cycling or severe premenstrual syndrome that could interfere with accurate assessment of the treatment effect
* History of substance abuse/dependence with less than one year remission
* GAF < 50
* Light treatment in the previous month
* Pregnant or lactating
* Antidepressant medications in the previous month
* Nightwork or other habitual alteration of sleep/wake cycle
* Medical conditions that affect mood or produce hallmark symptoms of mood disorder
* Use of photosensitizing medications (amiodarone, benoxaprofen, chlorpromazine, demeclocycline, fleroxacin, nalidixic acid, ofloxacin, piroxicam, porfimer, psoralens, quinidine, temoporfin) or remedies (St. John's wort)
* Macular degeneration or cataract

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 24
Dates: Start 2005-05

PRIMARY OUTCOMES:
score on depression rating scale at weeks 1, 2, and 3 by rater blind to treatment condition

SECONDARY OUTCOMES:
score on hypomania/mania rating scale at weeks 1, 2, and 3
adverse effects reported to rater blind to treatment condition

CONTACTS AND LOCATIONS:
Overall Officials: Janis L Anderson, Ph.D, Principal Investigator — Brigham and Women's Hospital
Locations (1):
- SAD Clinical Services, BWH Psychiatry; 221 Longwood Ave., Boston, Massachusetts, United States

REFERENCES:
- [Derived] Anderson JL, Glod CA, Dai J, Cao Y, Lockley SW. Lux vs. wavelength in light treatment of Seasonal Affective Disorder. Acta Psychiatr Scand. 2009 Sep;120(3):203-12. doi: 10.1111/j.1600-0447.2009.01345.x. Epub 2009 Feb 3. PMID 19207131
- See also: study announcement — http://www.brighamandwomens.org/psychiatry/Research/sadresearch.aspx